CLINICAL TRIAL: NCT06161792
Title: A Randomized, Placebo-Controlled, Double-Blind, Parallel, Phase 2 Study to Evaluate the Efficacy and Safety of RCN3028 in Treatment of Drug-Induced Moderate to Severe Vasomotor Symptoms in Breast Cancer Subjects
Brief Title: Evaluate RCN3028 in Treatment of Drug-Induced VMS in Breast Cancer
Acronym: VMS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Difficulty in recruiting breast cancer patients, leading to a slow rate of case enrollment.
Sponsor: Yung Shin Pharm. Ind. Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: YSP-RCN3028-03
Record Dates: First submitted 2023-10-23; First posted 2023-12-08 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-11

CONDITIONS: Hot Flashes; Breast Cancer
Keywords: Hot Flashes
MeSH Terms: conditions — Hot Flashes; Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- I placebo capsule (Placebo Comparator): Subjects will be enrolled to about 14-days of placebo-run-in period.
  Other Names:
  RCN3028 placebo
  Interventions: Drug: Placebo
- II RCN3028 0.8 mg capsule (Experimental): Subjects will be enrolled to about 14-days of placebo-run-in period. Treatment started at 0.4 mg, titrated to 0.8 mg for maintenance phase.
  Other Names:
  RCN3028 0.8 mg capsule
  Interventions: Drug: 0.8 mg RCN3028

INTERVENTIONS:
Drug: 0.8 mg RCN3028 — Oral
  Arms: II RCN3028 0.8 mg capsule
Drug: Placebo — Oral
  Arms: I placebo capsule

SUMMARY:
Due to the fact that majority of breast cancers are estrogen-receptor and/or progesterone receptor positive, tamoxifen and aromatase inhibitors (AIs) are among the mainstay therapies to treat breast cancer. Prior clinical studies of tamoxifen suggested that up to 80 % of patients experienced hot flashes during therapy with tamoxifen, and 30 % defined their symptoms as severe. Despite the high efficacy of tamoxifen, the harmful side effects have been identified in previous studies as a significant reason for not persisting with the treatment in 16 - 30 % of breast cancer patients.

The primary purpose of this study is to determine if RCN3028 is effective and safe in the treatment of moderate to severe vasomotor symptoms associated. In accordance with the latest FDA guidance study participants will have a minimum of 7 moderate to sever hot flashes per day, or 50 per week at baseline.

DETAILED DESCRIPTION:
Hot flashes are the most common symptom of menopause and affect almost 75% of menopausal women. Clinical evidence indicates potent antagonists of 5-HT2a are more likely to cause hypothermia. Risperidone is a potent 5-HT2a and a dopamine D2 receptor antagonist and is proposed to have effect on reduction of hot flashes through its dopaminergic and serotonergic antagonism.

Breast cancer is one of the most common cancers in women, according to the cancer registration report of the Ministry of Health and Welfare (MOHW), in 2014, up to 11,976 women suffered from breast cancer, which meant 33 women suffered from breast cancer daily. Recent epidemiology further disclosed that the incidence of breast cancer was top-ranked (70.74 per 100,000) among cancers of Taiwanese women in 2014.

Due to the fact that majority of breast cancers are estrogen-receptor and/or progesterone receptor positive, tamoxifen and aromatase inhibitors (AIs) are among the mainstay therapies to treat breast cancer. Prior clinical studies of tamoxifen suggested that up to 80 % of patients experienced hot flashes during therapy with tamoxifen, and 30 % defined their symptoms as severe. Despite the high efficacy of tamoxifen, the harmful side effects have been identified in previous studies as a significant reason for not persisting with the treatment in 16 - 30 % of breast cancer patients.

The primary purpose of this study is to determine if RCN3028 is effective and safe in the treatment of moderate to severe vasomotor symptoms associated. In accordance with the latest FDA guidance study participants will have a minimum of 7 moderate to sever hot flashes per day, or 50 per week at baseline.

With recent advances of treatment modalities, more than 80% of women with a newly diagnosed breast cancer are expected to survive their disease for 5 years or more. One of the most common complaints was hot flashes induced by the treatment of breast cancer (i.e., tamoxifen induced hot flashes).

In general, hormone replacement therapy (HRT) is the most effective treatment for VMS (hot flashes). However, HRT has been associated with increased risk of recurrence in breast cancer survivors . Moreover, there is some evidence that HRT may not be as effective in women using tamoxifen. Therefore, a new therapy for treating hot flashes in breast cancer patients without increasing the risk of cancer recurrence is needed for such patient population, for example, a non-hormonal therapy. FDA approved low-dose paroxetine capsules (Brisdelle®) as a non-hormonal therapy for the treatment of moderate-to-severe vasomotor symptoms associated with menopause, despite the modest efficacy as compared with placebo, suicidal ideation and the drug-drug interactions (i.e., Brisdelle® and tamoxifen) . Brisdelle® itself is an antidepressant of selective serotonin reuptake inhibitors (SSRI) class. Several trials have recently demonstrated a role for SSRIs and serotonin-norepinephrine reuptake inhibitors (SNRIs) for the treatment of VMS.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects (aged 20 years or order) with confirmed diagnosis of breast cancer who have completed chemotherapy and radiotherapy, and are on a stable dose of tamoxifen or aromatase inhibitors (AIs) for at least 8 weeks at baseline and will maintain the same treatment regimen and dose throughout the study.
* Reported 7 or more moderate to severe hot flashes per day (average) or 50 moderate to severe hot flashes per week at baseline.
* Screening laboratory values for hematopoietic, hepatic, and renal functions are within the following ranges:

  * Hematopoietic : Absolute neutrophil count ≥ 1,500/mm3、Platelet count ≥ 100,000/mm3
  * Hepatic : Glutamic Oxaloacetic Transaminase/Glutamic Pyruvic Transaminase ≤ 3 times upper limit of normal (ULN)、Bilirubin ≤ 1.5 times ULN
  * Renal : Creatinine ≤ 1.5 times ULN
* Having Eastern Collaborative Oncology Group (ECOG) Performance Status of ≤ 1.
* Ability to understand and follow the instructions of the investigator, including completion of the study procedures as described in the protocol (i.e., VMS episode event log).
* Able and willing to provide written informed consent.

Exclusion Criteria:

* Subjects are pregnant or breastfeeding.
* Female subjects who have childbearing potential, but they are not willing to use effective contraceptive methods during study period and for 1 week afterward.
* Subjects who have multiple primary cancers (except for completely resected basal cell cancer, stage I squamous cell carcinoma, carcinoma in situ, intramucosal carcinoma, or superficial bladder cancer or any other cancer from which the patient has been recurrence-free for at least 5 years).
* Subjects who have inoperable breast cancer (Stage IIIB/IIIC/IV).
* Subjects who have the following medical history: myocardial infarction, congestive heart failure, significant ischemic or valvular heart disease, clinically active interstitial lung disease.
* Subjects who have systolic blood pressure (BP) outside the range 100 to 150 mmHg, diastolic BP outside the range 60 to 90 mmHg, and/or heart rate outside the range 50 to 100 bpm at baseline.
* Subjects who had received treatment for hypotension within 30 days prior to screening visit.
* Subjects who have uncontrolled hyperglycemia, HbA1c ≥ 7% at baseline.
* Subjects who have clinical significant conditions such as acute myocardial infarction or stroke with 6 months of randomization.
* Subjects who have a history of Parkinson's disease.
* Subjects are taking risperidone in the 30 days prior to screening visit.
* Subjects who had participated in another clinical trial and received an investigational drug within 30 days prior to screening visit.
* Subjects having a known history of allergic reaction, hypersensitivity or clinically significant intolerance to ingredients of the study drug.
* Subjects with a current drug or alcohol abuse problem as judged by the investigator.
* Subjects who are considered unreliable as to medication compliance or adherence to scheduled appointments or for other reasons are felt to be inappropriate for inclusion in the study as determined by the investigators.
* Subjects who use Selective Serotonin Reuptake Inhibitors (SSRI) or Serotonin-Norepinephrine Reuptake Inhibitors (SNRI), within 4 weeks prior to screening visit.
* Subjects who use herbal or dietary supplements, including black cohosh, soy, phytoestrogens or over the counter agents known to possibly be effective for the treatment of vasomotor symptoms within 2 weeks prior to baseline.
* Subjects who have serious, unstable, or clinically significant medical or psychological conditions, which, in the opinion of the investigator(s), would compromise the subject's participation in the study.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-11-07 (Actual); Primary Completion 2022-03-14 (Actual); Study Completion 2022-04-20 (Actual)

PRIMARY OUTCOMES:
Mean change in frequency of moderate to severe VMS | 4, 12 weeks
  Mean change in frequency numbers of moderate to severe VMS(Vasomotor Symptoms) from baseline to weeks 4 and week 12. The VMS episode event log recorded the frequency of hot flashes per day, such mild, moderate, severe, nighttime awakening number.
Mean change in severity of moderate to severe VMS | 4, 12 weeks
  Mean change in severity score of moderate to severe VMS from baseline to weeks 4 and week 12. The severity score for VMS for each subject is calculated as the sum of 2 times the number of moderate VMS, plus 3 times the number of severe VMS, divided by the total number of moderate and severe VMS.

SECONDARY OUTCOMES:
Menopause Specific Quality of Life Questionnaire | 12 weeks
  Menopause Specific Quality of Life Questionnaire will be completed at baseline, week 4, week 8 and week 12. Score on a scale Menopause Specific Quality of Life (MENQOL) questionnaire 0=not bothered at all - 6=extremely bothered. 4 domains, mean calculated for set of questions in each domain.
The 50%, 75% and 100% responder rates | 12 weeks
  Subject who had a reduction in the number of moderate and severe hot flashes of at least 50%, at least 75% and 100% from baseline.
The time to onset of efficacy | 12 weeks
  50% reduction in hot flashes for at least 3 consecutive days. The duration of first treatment used to first onset on efficacy will be calculated.
Subject's and Physician's Global Assessment | 12 weeks
  At the end of treatment Visit (week 12) each subject will provide an overall evaluation of study treatment by completing a Subject's Global Assessment. The rating scale for the final assessment by the subject includes: much worse, worse, unchanged, improved, much improved or free of symptoms. At week 12 each investigator will be asked to rate their subject's response to therapy using the same scale.
Frequencies(number and percentage) of subjects with treatment-emergent AEs (TEAEs) | 12 weeks
  Frequencies (number and percentage) of subjects with one or more treatment-emergent AEs (TEAEs) will be summarized by treatment arm, by the Medical Dictionary for Regulatory Activities (MedDRA) system with respect to System Organ Class (SOC) and preferred term.
Change from baseline in weekly weighted severity score. | 12 weeks
  calculated for each week as 2 times the number of moderate hot flashes plus 3 times the number of severe hot flashes plus 3 times the number of nighttime awakenings.
  The severity of VMS is defined as follows:
  1. Mild: sensation of heat without sweating;
  2. Moderate: sensation of heat with sweating, able to continue activity;
  3. Severe: sensation of heat with sweating, causing cessation of activity.
  4. Nighttime awakenings (i.e., episodes that wake the patient from sleep) associated with hot flashes are recorded separately and are considered severe.
Change from baseline in the number of mild, moderate, and severe hot flashes. | 12 weeks
  The weekly frequency will be calculated for each visit.
Change from baseline in the number of nighttime awakenings because of hot flashes. | 12 weeks
  The weekly frequency will be calculated for each visit.

CONTACTS AND LOCATIONS:
Overall Officials: hui-Ling Shieh, PhD, Study Director — Yung Shin Pharm. Ind. Co., Ltd.
Locations (4):
- Taiwan (4):
  - Changhua Christain Hospital, Changhua
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Taipei Medical University Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No